CLINICAL TRIAL: NCT02845232
Title: Economic Analysis of Blood Product Transfusions According to the Treatment of Acute Myeloid Leukaemia in the Elderly
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0461
Record Dates: First submitted 2016-07-20; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Therapy; Blood transfusion; Cost-effectiveness; Prognosis
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Intensive chemotherapy: First group: 68 patients receiving a combination of intermediate-dose cytarabine and an anthracycline. One patient with acute promyelocytic leukaemia (APL) also received all-trans retinoic acid (ATRA).
  Interventions: Other: Transfusion
- Lower-intensity treatments: The second study group comprised 70 patients who were treated on frontline by lower-intensity treatments [LD-AraC(39 patients), azacitidine (16 patients), decitabine (11 patients),tipifarnib (3 patients), or ATRA (1 patient)]. Patients received LD-AraC 20 mg once or twice daily (according to physician'schoice) by subcutaneous injection for 10 consecutive days. Azacitidine was given at the dose of 75 mg/m2/day for 7 consecutive days by sc injection. Decitabine was administered by intravenous route once daily at 20 mg/m2 for 5 consecutive days. Tipifarnib was given at 600 mg administered orally twice daily for 21 consecutive days in 4-week cycles. ATRA was given at 45 mg/m2until CR achievement followed by maintenance combining 6-mercaptopurine with methotrexate.
  Interventions: Other: Transfusion
- Best Supportive Care: The last study group comprises 76 patients: 31 patients received supportive care, while 36 patients also received hydroxyurea and 9 patients received 6-mercaptopurine.
  Interventions: Other: Transfusion

INTERVENTIONS:
Other: Transfusion — The number and type of blood products administered were registered from the time of diagnosis to the time of death corresponding for all patients to the time of last follow-up. Transfusion of a single unit of packed red blood cell (PRBC) or one whole blood-derived platelet concentrate (PC) or fresh frozen plasma (FFP) was considered a transfusion event and considered for statistical analysis.

SUMMARY:
Blood transfusion requirement represents one of the most significant cost driver associated with acute myeloid leukemia (AML). In addition to an increase prevalence of co morbidities in older patients, AML in older patients is more often associated with adverse features than in younger adults. Physicians might therefore decide to offer palliative or supportive care rather than intensive chemotherapy. An alternative treatment could be low-intensity therapy, such as LD-AraC or hypomethylating agents, which demonstrated better results than only Best Supportive care (BSC). Blood transfusion requirement represents one of the most significant cost driver associated with AML.

The present study assesses the cost-effectiveness of intensive chemotherapy versus Best Supportive Care (BSC) versus alternative therapies (hypomethylating agents, low-dose cytosine arabinoside (LD-AraC), or other investigational drugs) in elderly patients aged 70 years or older regarding blood product transfusions from a French payer perspective. Intensive chemotherapy and BSC were the comparators in this analysis, since they continue to represent the most commonly used treatment for elderly AML according to the defined status of patients considered as 'fit' or 'unfit' for intensive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years old
* AML according to the World Health Organization (WHO) criteria (% of blasts ≥ 20% in bone marrow aspiration).
* All FAB subtypes.
* Any type of AML (de novo or secondary)
* All participants to clinical trials gave their written informed consent

Exclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) score ≥2
* Active uncontrolled infection

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Three groups of elderly patients aged 70 years or older, with AML. First group: 68 patients receiving a combination of intermediate-dose cytarabine and an anthracycline. One patient with acute promyelocytic leukaemia (APL) also received all-trans retinoic acid (ATRA).
  The second study group comprised 70 patients who were treated on frontline by lower-intensity treatments [LD-AraC(39 patients), azacitidine (16 patients), decitabine (11 patients),tipifarnib (3 patients), or ATRA (1 patient)].
  The last study group comprises 76 patients: 31 patients received supportive care, while 36 patients also received hydroxyurea and 9 patients received 6-mercaptopurine.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Estimation of mean blood product transfusions costs (in euros) per patient according to overall survival | From starting treatment to death from any cause (up to 21 months)
  The cost-effectiveness of blood product transfusion was determined among initial treatment subgroups: patients receiving intensive chemotherapy, patients receiving low-intensity treatments, and patients treated only by BSC.

SECONDARY OUTCOMES:
Complete remission (CR) rate | Duration of study (Month 21)
  Complete remission (CR) was defined by bone marrow aspiration, which was required to consist of more than 50% normal cellularity with evidence of trilineage maturation and less than 5% bone marrow blasts, no evidence of extramedullary disease, and regeneration of the peripheral neutrophil count to 1.0 × 109/L and the platelet count to 100 × 109/L. The persistence of myelodysplastic features did not exclude the diagnosis of CR.
Number of blood product transfusions per patient | Duration of study (Month 21)
  Decisions concerning transfusion indications were based on institutional policy and the clinical judgment of treating physicians. Transfusion practice was consistent during the period of study. Prophylactic transfusions were consistently given at morning platelet counts of < 20 ×109/L and haemoglobin level < 80 g/L. Protocol Blood products were leukoreduced through discarding the buffy coat and administered through a standard 140 to 170 µm blood filter but were not irradiated

CONTACTS AND LOCATIONS:
Overall Officials: Xavier THOMAS, MD-PhD, Principal Investigator — Hospices Civils de Lyon - Centre Hospitalier Lyon Sud
Locations (1):
- Hospices Civils de Lyon - Centre Hospitalier Lyon Sud, 165 Chemin du Grand Revoyet, Pierre-Bénite, France